CLINICAL TRIAL: NCT01915706
Title: The Effect of Scheduled Ripcord Removal on the Outcomes of Baerveldt 350 Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00047845
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Glaucoma
Keywords: Glaucoma drainage device; Baerveldt 350; Ripcord; Complications
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (No Intervention): Patients randomized to observation will be observed during the post-operative period for spontaneous Baerveldt-350 tube opening. The ripcord will not be removed unless deemed medically necessary by the study physician.
- Ripcord removal (Experimental): Patients randomized to intervention will have their ripcords removed in clinic at post-operative week 3.
  Interventions: Procedure: Ripcord removal

INTERVENTIONS:
Procedure: Ripcord removal — Patients randomized to intervention will have their ripcords removed in clinic at post-operative week 3. Ripcord removal will be performed by study PI at the slit lamp with standard of care sterile technique and topical/local anesthesia. Patients will be monitored 30 minutes following ripcord removal for intraocular pressure as well as complications.
  Arms: Ripcord removal

SUMMARY:
The purpose of this study is to compare the post-operative complication rates and surgical outcomes in patients with a Baerveldt 350 implant following scheduled rip-cord removal in clinic at post-operative week 3 versus spontaneous tube opening. Patients age 18 or greater with uncontrolled glaucoma and scheduled to undergo their first superotemporal Baerveldt 350 implant will be recruited and randomized at the time of enrollment to either scheduled ripcord removal at post-operative week 3 or no ripcord removal. Incidence of complications will be documented and compared between the 2 groups. The final intraocular pressure control between the 2 groups will also be compared in a secondary outcome analysis. This study will help to establish post-operative management guidelines to minimize complications and improve intraocular pressure lowering success following Baerveldt 350 implantation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older at screening. There is no upper age limit.
* Inadequately controlled glaucoma refractory to maximum therapy
* Suitable candidate for Baerveldt-350 implant in the superotemporal quadrant in the study eye, which the physician deems as medically necessary.
* Capable and willing to provide consent

Exclusion Criteria:

* Unable or unwilling to provide consent
* Any previous ocular surgery other than cataract extraction or trabeculectomy
* Any previous ocular surgeries in the study eye preventing placement of the Baerveldt-350 implant in the superotemporal quadrant
* Any abnormality other than glaucoma in the study eye that could affect tonometry.
* Presence or history of any abnormality or disorder that could interfere with the study procedure or prevent the successful completion of the study.
* Monocularity (where best corrected visual acuity in the non-operative eye is worse than 20/200)
* Any significant unstable cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Known pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09; Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative complications | Up to 6 months
  Incidence of complications (including but not limited to shallowing of the anterior chamber, hypotony, choroidal effusion and choroidal hemorrhage) will be documented and compared between the 2 groups.

SECONDARY OUTCOMES:
Incidence of successful intraocular pressure control | Post-operative month 6
  Final intraocular pressure at post-operative month 6 will be assessed and incidence of successful intraocular pressure control will be compared. Successful intraocular pressure control is defined as unqualified when the intraocular pressure is between 6 and 18 mmHg or a 25% reduction from the pre-surgical intraocular pressure without medication and qualified when pressure-lowering therapies are required to maintain intraocular pressure at that level.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Herndon, M.D., Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] An SJ, Wen JC, Quist MS, Mathenge EW, Vin A, Herndon LW. Scheduled Postoperative Ripcord Removal in Baerveldt 350 Implants: A Prospective, Randomized Trial. J Glaucoma. 2019 Feb;28(2):165-171. doi: 10.1097/IJG.0000000000001133. PMID 30689608